CLINICAL TRIAL: NCT03656081
Title: Therapeutic Efficacy Comparison of a Six-month Treatment by Itraconazole and Nebulised Ambisome® Versus Treatment by Itraconazole Alone in Non- or Mildly- Immunocompromised Patients with Chronic Pulmonary Aspergillosis: a Prospective, Randomized, Single Blind Study, (single Aspergilloma Excluded)
Brief Title: Chronic Pulmonary Aspergillosis and Ambisome Aerosol with Itraconazole
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPAAARI
Record Dates: First submitted 2018-07-19; First posted 2018-09-04 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pulmonary Aspergillosis
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Itraconazole & inhaled placebo (Placebo Comparator): Itraconazole 200 mg x 2/day associated with inactive nebulised treatment (isotonic saline) twice a week during 24 weeks.
  Interventions: Drug: inhaled placebo; Drug: Itraconazole
- Itraconazole & inhaled Ambisome® (Experimental): Itraconazole 200 mg x 2/day associated with inhaled liposomal amphotericin B (Ambisome®) at 25 mg twice a week during 24 weeks
  Interventions: Drug: inhaled Ambisome®; Drug: Itraconazole

INTERVENTIONS:
Drug: inhaled Ambisome® — inhaled liposomal amphotericin B = inhaled LAmB
  Arms: Itraconazole & inhaled Ambisome®
Drug: inhaled placebo — inhaled isotonic saline
  Other Names: placebo (for Ambisome®)
  Arms: Itraconazole & inhaled placebo
Drug: Itraconazole — Itraconazole tablet
  Other Names: Sporanox®

SUMMARY:
This study compares the therapeutic (clinical and radiological) efficacy of a six-month treatment by itraconazole and nebulised Ambisome® (liposomal amphotericin B = LAmB) versus treatment by itraconazole alone, in non - or mildly - immunocompromised patients affected by Chronic Pulmonary Aspergillosis (single aspergilloma excluded).

• Control arm: Itraconazole 200 mg x 2/day associated with inactive nebulised treatment twice a week during 24 weeks.

• Experimental arm: Itraconazole 200 mg x 2/day associated with nebulised LAmB, at 25 mg twice a week during 24 weeks.

Follow up duration for the patients will be 24 months (12 months minimum) after discontinuation of the treatment being studied.

ELIGIBILITY:
Inclusion Criteria:

All adult patients affected with Chronic Pulmonary Aspergillosis (CPA) "de novo" or in relapse (without any history of resistance to itraconazole) combining the following criteria are eligible:

1. Patient with an Aspergillus bronchopulmonary infection, be it cavitary, fibrotic, necrotizing (SIA/Semi Invasive Aspergillosis) or nodular and documented by compatible thoracic CT-scan images ;
2. Associated with one of the following criteria:

   * positive detection of anti-Aspergillus IgG and/or precipitating anti-aspergillus antibodies, according to the positivity threshold of the laboratory performing the technique,
   * positive direct examination of Aspergillus or positive culture, from bronchopulmonary samples (expectoration or endoscopic aspiration),
   * revealing aspergillar hyphae/filaments on histological samples
3. Men or women age ≥ 18 years;
4. For the women of childbearing age: women having a negative serum pregnancy test, having a contraception highly effective and accepting to pursue it during at least the first 12 months of the study;
5. Patient legally free and not subject to any custody, guardianship, tutelage or subordination measures;
6. Participants must be affiliated to France's Health Care Regime (" Sécurité Sociale ");
7. Free and informed consent signed by each participating patient.

Exclusion Criteria:

1. - Patient affected with single aspergilloma
2. - Patient presenting a contraindication to itraconazole (including all contraindicated co-administrated medications as listed in the itraconazole SmPc, including notably medications with potential to prolong theQT interval)
3. - Patient presenting a contraindication to voriconazole and posaconazole (including all contraindicated coadministrated medications as listed in the SmPc)
4. - Intolerance to beta2-agonists
5. - Notion of relapse with isolation of an Aspergillus resistant to itraconazole
6. - History of hypersensitivity reaction to liposomal amphotericin B or to itraconazole or to any other constituent
7. - Patient having presented complications related to a previous treatment by nebulised LAmB
8. - Patient received an oral (excepted oral Amphotericin B), parenteral or intra-cavity antifungal treatment within the last 2 months
9. - Severe renal failure (clearance <30 ml / min).
10. - Hepatic failure with transaminase and alkaline phosphatase values > 5 times normal
11. - Significant abnormality of the blood cell and platelet counts (at the discretion of the investigator)
12. - Concomitant use of one or several of treatments contra-indicated with the experimental or non-experimental treatment
13. - Ventricular dysfunction such as congestive cardiac failure or history of congestive cardiac failure or patients with risk(s) factors of cardiac arrhythmia or symptomatic arrhythmia with a prolongation of the corrected QT interval > 450 msec in men and 470 msec in women or treated by medication known to prolong QT interval, or prolongation of the corrected QT interval > 450 msec in men and 470 msec in women.
14. - Invasive pulmonary Aspergillosis, Allergic Bronchopulmonary Aspergillosis
15. - Chronic Pulmonary Aspergillosis with indication for surgical intervention within 6 months from the start
16. - Patients with Cystic Fibrosis
17. - Immunocompromised patients
18. - Threatening hemoptysis, with impossibility to defer surgical procedures (but patients contraindicated to surgery may be included after resolution of the hemoptysis)
19. - Tuberculosis or progressive non-tuberculous mycobacteria
20. - Respiratory infection aggravating the underlying CPA (patient may be included after eradication of infection)
21. - Patient refusing to participate
22. - Protected majors in the meaning of the law, non affiliated persons or with no social security scheme, persons deprived of liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and finally patients in emergencies.
23. - Patient in exclusion period following participation in another interventional study evaluating antifungals or medicines
24. - Women at age to procreate and not using highly effective contraception, pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Composite efficacy criterion defined by the association of clinical improvement/stability and radiological improvement evaluated at 6 months | 6 months
  • Clinical improvement or stability is evaluated using the Respiratory Symptom Score based on 6 items (cough, expectoration, dyspnea, hemoptysis, chest pain, and nocturnal awakening ) quoted with a 10 cm visual analogical scale).
  Stability is defined by a score variation between -25 and +25%, while improvement is defined by a decrease in score greater than 25%.
  • Radiological improvement is based on the analysis of CT-scan parameters (a committee consisting on two chest radiologists wil perform centrally and parallel analyses of each CT-scan blinded to the study treatment allocation to reach a final decision by consensus)
  The radiological improvement (binary variable) is defined by a consensual score based on the evolution of the various radiological parameters (cavity, fungus ball, alveolar condensation, nodules) according to validated thresholds.

SECONDARY OUTCOMES:
major events during follow-up period | month 6 to month 30
relapse | month 6 to month 30
mycological response | after 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cendrine GODET, MD, Principal Investigator — Bichat Hospital, AP-HP
Locations (1):
- CHU Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No